CLINICAL TRIAL: NCT05332444
Title: Efficacies of Susceptibility-guided vs Empiric Therapy for Rescue Treatment of Helicobacter Pylori Infection - A Prospective Randomized, Comparative Study
Brief Title: Efficacies of Susceptibility-guided vs Empiric Therapy for Rescue Treatment of Helicobacter Pylori Infection
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 202112229MINB
Record Dates: First submitted 2022-04-10; First posted 2022-04-18 (Actual); Last update posted 2025-09-23 (Actual); Status verified 2025-09

CONDITIONS: Helicobacter Pylori Infection
Keywords: Helicobacter pylori; antimicrobial susceptibility testing; minimal inhibitory concentration; susceptibility-guided tailored therapy; guideline-recommended empiric therapy
MeSH Terms: interventions — Rabeprazole; Amoxicillin; Clarithromycin; Levofloxacin; Metronidazole; Tetracycline

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- susceptibility-guided tailored therapy (Group A) (Experimental): Includes 5 treatment options. The priority order of treatment regimens is based on the selection principal through AST with MIC profile.
  1. clarithromycin triple therapy: include rabeprazole 20mg bid, amoxicillin 1 g bid, and clarithromycin 500 mg bid, for 14 days; or 2. levofloxacin triple therapy: include rapeprazole 20 mg bid, amoxicillin 1 g bid, and levofloxacin 500 mg bid, for 14 days; or 3. metronidazole triple therapy: include rabeprazole 20 mg bid, amoxicillin 500 mg qid, and metronidazole 250 mg qid, for 14 days; or 4. high-dose dual therapy: include rabeprazole 20 mg qid, amoxicillin 750 mg qid, for 14 days; or 5. bismuth quadruple therapy: include rabeprazole 20 mg bid, bismuth 120 mg qid, metronidazole 500 mg tid, and tetracycline 500 mg qid, for 14 days.
  Interventions: Drug: susceptibility-guided tailored therapy (Group A)
- guidelines-recommended empiric therapy (Group B) (Active Comparator): bismuth quadruple therapy: include rabeprazole 20 mg bid, bismuth 120 mg qid, metronidazole 500 mg tid, and tetracycline 500 mg qid, for 14 days.
  Interventions: Drug: guidelines-recommended empiric therapy (Group B)

INTERVENTIONS:
Drug: susceptibility-guided tailored therapy (Group A) — Includes 5 treatment options. The priority order of treatment regimens is based on the selection principal through AST with MIC profile.
  1. clarithromycin triple therapy: include rabeprazole 20mg bid, amoxicillin 1 g bid, and clarithromycin 500 mg bid, for 14 days; or 2. levofloxacin triple therapy: include rapeprazole 20 mg bid, amoxicillin 1 g bid, and levofloxacin 500 mg bid, for 14 days; or 3. metronidazole triple therapy: include rabeprazole 20 mg bid, amoxicillin 500 mg qid, and metronidazole 250 mg qid, for 14 days; or 4. high-dose dual therapy: include rabeprazole 20 mg qid, amoxicillin 750 mg qid, for 14 days; or 5. bismuth quadruple therapy: include rabeprazole 20 mg bid, bismuth 120 mg qid, metronidazole 500 mg tid, and tetracycline 500 mg qid, for 14 days.
  Other Names: Proton pump inhibitor: Rabeprazole, Pariet®; Antibiotics: Amoxicillin, Amoxicillin®; Clarithromycin, Klaricid®; Levofloxacin, Cravit®; Metronidazole, Metrozole®; Tetracyclline, tetracycline®; Colloidal Bismuth: Tripotassium dicitrate bismuthate, KCB®
  Arms: susceptibility-guided tailored therapy (Group A)
Drug: guidelines-recommended empiric therapy (Group B) — bismuth quadruple therapy: include rabeprazole 20 mg bid, bismuth 120 mg qid, metronidazole 500 mg tid, and tetracycline 500 mg qid, for 14 days.
  Other Names: Proton pump inhibitor: Rabeprazole, Pariet®; Antibiotics: Metronidazole, Metrozole®; Tetracyclline, tetracycline®; Colloidal Bismuth: Tripotassium dicitrate bismuthate, KCB®
  Arms: guidelines-recommended empiric therapy (Group B)

SUMMARY:
The prevalence of H. pylori antibiotic resistance has reached an alarming level worldwide. Antibiotic stewardship programs should be urgently developed and implemented. However, H. pylori antimicrobial susceptibility testing (AST) is rarely offered, making local resistance patterns not easily available. Guideline-recommended empiric therapies (GR-ET) may no longer reliably achieve high cure rate in the era of increasing antibiotic resistance. susceptibility-guided tailored therapy (SG-TT) may be a good choice to solve this problem.

The aims of this study are:

1. to compare the efficacy of SG-TT with GR-ET as rescue regimens for H. pylori eradication;
2. to compare the patient adherence and adverse effects of these treatment regimens;
3. to investigate factors that may influence H. pylori eradication by these treatment regimens.

DETAILED DESCRIPTION:
This prospective multicenter randomized comparative study will be conducted at the National Taiwan University Hospital, NTUH Bei-Hu Branch, NTUH Hsin-Chu Branch, Taipei City Hospital Renai Branch, Buddhist Tzu Chi General Hospital, and Mennonite Christian Hospital in Hualien. The study protocol will be approved by the independent ethics boards or committees of each hospital. Patients, aged >= 20, having H. pylori-positive chronic gastritis with/without peptic ulcers (duodenal or gastric ulcers) will be recruited. If the patients failed anti-H. pylori therapy previously, these patients will be invited to enter this study for evaluating the efficacy of these rescue regimens.

A computed generated random numbers sequence will be blocked (1:1; block size 6) into two subgroups, say A, and B. After giving written informed consent, each patient will be randomly allocated, to one of two treatment groups:

group A - SG-TT (susceptibility-guided tailored therapy) : treated with 1. clarithromycin triple therapy, or 2. levofloxacin triple therapy, or 3. metronidazole triple therapy, or 4. high-dose dual therapy, or 5. bismuth quadruple therapy, by priority order base on the selection principal through AST with MIC profile;

group B -GR-ET (guidelines-recommended empiric therapy): treated with bismuth quadruple therapy.

All patients will be asked to complete a questionnaire and to record symptoms and drug consumption, and diet content daily during the treatment period. Post-treatment, the patients will be followed up at the Outpatients Clinic to investigate patient adherence and adverse effects of treatment. Four to eight weeks after termination of treatment, H. pylori infection status will be examined by the 13C-urea breath test (UBT). The CYP2C19 genotype of each participant will be analyzed by the polymerase chain reaction-based restriction fragment length polymorphism (PCR-RFLP) method.

ELIGIBILITY:
Inclusion Criteria:

Patients, aged >= 20, having H. pylori-positive chronic gastritis with/without peptic ulcers (duodenal or gastric ulcers) will be recruited. If the patients failed anti-H. pylori therapy previously, they will be invited to enter this study for evaluating the efficacy of these rescue regimens.

Exclusion Criteria:

1. pregnant or nursing woman;
2. serious concomitant illness and malignant tumor of any kind;
3. history of hypersensitivity to test drugs；
4. serious bleeding during the course of this ulcer;
5. previous gastric surgery;
6. receiving bismuth salts, PPIs, or antibiotics in the previous month.

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 450 (Estimated)
Dates: Start 2022-04-11 (Actual); Primary Completion 2025-09 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
to compare the eradication rate of SG-TT with GR-ET as rescue regimens for H. pylori eradication. | 3.5 years
  The eradication rate (efficacy) of these regimens will be evaluated by the result of C13-UBT in intention-to treat (ITT) and per-protocol (PP) analysis.

SECONDARY OUTCOMES:
to compare the patient adherence and frequency of adverse effects of these treatment regimens | 3.5 years
  The frequency of adverse events will be evaluated by the number of participant with adverse events and patient adherence will be evaluated by counting unused medication after the treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Jyh-Chin Yang, M.D.Ph.D., Principal Investigator — National Taiwan University Hospital
Locations (1):
- National Taiwan University Hospital, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: No